CLINICAL TRIAL: NCT03546075
Title: The Impact of Acute Trans-resveratrol Administration on Whole Body Metabolism During Cognitive Task Performance: a Double Blind, Randomised, Placebo-controlled Investigation.
Brief Title: The Impact of Acute Trans-resveratrol Administration on Whole Body Metabolism During Cognitive Demand.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Responsible Party: Principal Investigator, Tim Eschle, Principal investigator, Northumbria University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 42BB1
Record Dates: First submitted 2018-04-09; First posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Cognitive Change
Keywords: Cognition; Resveratrol; Whole body metabolism
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 500 mg Resveratrol (Experimental)
  Interventions: Dietary Supplement: Resveratrol
- 250 mg Resveratrol (Experimental)
  Interventions: Dietary Supplement: Resveratrol
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Resveratrol
  Arms: 250 mg Resveratrol; 500 mg Resveratrol
Other: Placebo
  Arms: Placebo

SUMMARY:
Background: Increased cerebral vaso-dilation during cognitive demand is hypothesised to improve cognitive performance due to an improved micronutrient status. Despite previous research demonstrating that oral resveratrol can modulate cerebral haemodynamics, this has not translated into expected improvements to cognitive performance in young, healthy populations. As the brain is the most metabolic organ in the body, even subtle changes to fuel utilization and overall energy expenditure are detectable during cognitive demand. The measurement of both overall energy expenditure and fuel utilization may provide further insight to the effects of resveratrol and whether oral supplementation of this polyphenol can provide clear, cognitive benefits in a young, healthy sample.

Objectives: The current study investigated the metabolic consequences of resveratrol on whole body metabolism and fuel oxidisation during cognitive performance.

Methods: This repeated measures, double blind, placebo controlled, balanced design required participants (N=24 for metabolic activity & N=26 for cognitive outcomes) to complete a serial subtraction demand battery at baseline, 45 minutes, 2 and 3 hours following 500 mg, 250 mg trans-resveratrol or inert placebo, on three separate occasions whilst connected to an on-line gas analysis system.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were able to give informed consent.
* Those who didn't meet any of the exclusion criteria.
* Those who took hormonal contraception (e.g. the pill, coil, implant, etc.) were still allowed to participate in the current study.

Exclusion Criteria:

* Participants who smoke.
* Participants below the age of 18 years or above 35 years at the time of giving consent to in role in the current study.
* Participants with Body Mass Index outside the range of 18-35 kg/m2.
* Participants with blood pressure greater than 140/90 HH/mg.
* Participants with a history of neurological, vascular or psychiatric illness (excluding depressive illness and anxiety).
* Participants with a current diagnosis of depression and / or anxiety.
* Participants with learning difficulties: dyslexia, dyscalculia or colour blindness.
* Participants with a visual impairment that cannot be corrected with glasses or contact lenses.
* Participants with frequent migraines that require medication (more than or equal to 1 per month).
* Participants with disorders of the blood.
* Participants with a heart disorder.
* Participants with diabetes.
* Participants with a respiratory disorder that requires regular medication (Note: asthma sufferers who only take their medication occasionally/as required were eligible for this study).
* Participants currently taking any prescription medications.
* Participants who have habitually used dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total).
* Participants with any food intolerances/sensitivities.
* Participants with a history of renal or hepatic disease, or other severe diseases of the gastrointestinal tract (e.g., iron accumulation, iron utilization disorders, hypercalcaemia, hypercalciuria), that are likely to interfere with metabolism/absorption/secretion of the product under investigation.
* Female participants who are currently pregnant, lactating or seeking to become pregnant.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2015-12-18 (Actual); Study Completion 2015-12-18 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 1 Hour
  Participants completed three Serial subtraction tasks (Serial 3, 7 & 17). Outcomes measured from all three of these tasks were the number correct entries and number of errors. The addition of the two outcomes can also provide a 'total' number of responses entered.
Whole body metabolism | 1 Hour
  Whole body energy expenditure was measured via indirect calorimetry and was reported in calories burned per minute (Kcal / min).
Fuel Oxidisation | 1 Hour
  Fuel oxidation was measured via indirect calorimetry and examined the rate of carbohydrate and fat oxidisation (both in grams per minute (g / min)).

SECONDARY OUTCOMES:
Pulmonary gases | 1 Hour
  An on-line gas analysis system was used to measure oxygen intake and carbon dioxide excretion (both in litres per minute (L / min)) from the participant's expired pulmonary air.